CLINICAL TRIAL: NCT06689514
Title: Study on the Effectiveness of Tranilast in the Treatment of Medium to Large Volume Benign Prostatic Hyperplasia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yifeng Jing (Other)
Responsible Party: Sponsor-Investigator, Yifeng Jing, Professor, Shanghai General Hospital, China
Organization: Shanghai General Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024HS197; 82270810 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Hypertrophy, Benign
Keywords: Prostatic Hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — tranilast

STUDY DESIGN:
Intervention Model Description: For patients who meet the inclusion criteria, the control group takes oral alpha receptor antagonists (according to the dosage specified in the instructions for treating BPH) (n=10); Low dose group: oral administration of 100mg TID of tranilast capsules (Qu Ke Shen, Yao Da Pharmaceutical)+oral administration of alpha receptor antagonist (according to the dosage specified in the instructions for treating BPH) (n=10); The high-dose group received oral administration of 200mg TID of tranilast capsules (Qu Ke Shen, Yao Da Pharmaceutical) and oral administration of alpha receptor antagonists (according to the instructions for treating BPH) (n=10). Take medication continuously for 6 months.
  This trial allows the combination of various drugs taken by patients for the treatment of hypertension, diabetes, hyperlipidemia and other chronic diseases, and allows the combination of antibiotics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Experimental)
  Interventions: Drug: alpha receptor antagonist
- Low dose group (Experimental)
  Interventions: Drug: alpha receptor antagonist; Drug: Low dose Tranilast
- High dose group (Experimental)
  Interventions: Drug: alpha receptor antagonist; Drug: High dose Tranilast

INTERVENTIONS:
Drug: alpha receptor antagonist — Oral administration of alpha receptor antagonist (according to the dosage specified in the instructions for treating BPH)
Drug: Low dose Tranilast — Oral administration of Tranilast Capsules (Qu Ke Shen, Yao Da Pharmaceutical) 100mg TID
  Arms: Low dose group
Drug: High dose Tranilast — Oral administration of Tranilast Capsules (Qu Ke Shen, Yao Da Pharmaceutical) 200mg TID
  Arms: High dose group

SUMMARY:
Benign prostatic hyperplasia (BPH) is one of the most common urinary and reproductive system diseases in elderly men. The preliminary research of the research group found that mast cells are cells that promote the progression of BPH, and the commonly used mast cell membrane stabilizer and TGF - β pathway inhibitor tranilast significantly inhibited the increase in prostate volume in animal experiments, which is considered to have potential applications in the treatment of BPH. This study plans to include 30 patients with medium to large volume BPH and experimentally explore the efficacy and safety of tranilast in the treatment of medium to large volume BPH.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is one of the most common urinary and reproductive system diseases in elderly men. The incidence of histological BPH in males aged 60 and above is over 50%, reaching as high as 83% at the age of 80. About 50% of BPH cases can lead to moderate to severe lower urinary tract symptoms (LUTS), and even serious complications such as hydronephrosis, which greatly affects the quality of life and health of patients, and also brings heavy social and medical burdens.

One of the important risk factors for the clinical progression of BPH is prostate volume. The risk of acute urinary retention and surgical intervention in BPH patients increased significantly with the increase of prostate volume. Medium to large volume prostate (prostate volume ≥ 60mL) is more likely to cause bladder outlet obstruction and severe hematuria, and surgical treatment is relatively difficult, with significantly increased surgical difficulty and complications. Therefore, controlling prostate volume is crucial in the treatment of benign prostatic hyperplasia.

At present, the commonly used drugs for the treatment of large volume prostate hyperplasia in clinical practice are 5 α - reductase inhibitors and α - receptor antagonists. The mechanism of action of 5 α - reductase inhibitors (such as finasteride, aprepit, etc.) is to inhibit the production of dihydrotestosterone to reduce prostate volume. However, about 40% of patients have poor reactions to these drugs, and long-term use of these drugs can lead to adverse reactions such as impaired sexual function (erectile dysfunction, decreased libido, etc.), breast discomfort, and rash. The mechanism of action of alpha receptor antagonists (such as doxazosin, tamsulosin, etc.) is to reduce urethral smooth muscle pressure and alleviate LUTS symptoms caused by BPH, but they cannot intervene in the continuous increase of prostate volume.

Quinilast is a highly effective and safe stabilizer for mast cells, TGF - β pathway inhibitor, and anti-inflammatory agent. It has a stabilizing effect on the cell membrane of mast cells and eosinophils, preventing their degranulation and inhibiting the release of histamine and 5-hydroxytryptamine allergens. It has a significant inhibitory effect on IgE antibody induced skin allergies and experimental asthma in rats. Quinilast can also inhibit collagen synthesis in fibroblasts and is currently widely used to treat allergic diseases and scars. After oral administration, the drug is rapidly absorbed in the gastrointestinal tract, with a peak plasma concentration time of 2-3 hours. It is widely distributed in all organs and tissues, with the highest concentration in the bronchi and lungs, followed by the liver, kidneys, and small intestine. The plasma half-life is 5-8.6 hours, and the blood drug concentration significantly decreases by 24 hours, making it difficult to detect after 48 hours. Metabolized in the liver, after administration, it is mainly excreted from the urine. Metabolites in the body include the demethylation product of tranilast at position 4, as well as the combination of sulfuric acid and glucuronic acid. Previous studies have confirmed that the TGF - β pathway is one of the important pathways that promote the occurrence and development of BPH. Our research confirms that the phenomenon of endothelial mesenchymal transition is an important factor in promoting the progression of BPH.

TGF - β 1 and VEGFA secreted by mast cells are important cytokines that promote endothelial mesenchymal transition in BPH, and stabilizing mast cells can inhibit endothelial cell to mesenchymal transition. The investigators confirmed through animal experiments that oral administration of tranilast (100mg/kg/d, n=10) to BPH mice for 30 consecutive days resulted in a decrease in endothelial mesenchymal transition and degree of BPH in the prostate of the mice. There was no statistically significant difference in body weight compared to the control group, and no mice died. Therefore, the investigators believe that tranilast has a promising application prospect in the treatment of BPH.

The commonly used dose of tranilast in clinical treatment of allergic diseases and scars is 100mg, three times a day (TID). There are currently no research reports on the use of tranilast for the treatment of BPH, so the effective dosage of tranilast for the treatment of BPH is not clear. Tranilast has carried out a long-term clinical trial (PRESTO test) for the treatment of atherosclerosis for more than 10000 people with a daily dose of 600mg and 900mg. The common adverse reactions (1% -10%) are nausea, abnormal liver function, and high serum creatinine. The adverse reactions will disappear after drug withdrawal. Based on our previous foundation, common dosages of tranilast, and considerations of dosage and safety in previous clinical trials, the investigators set up a low-dose group (tranilast 100mg TID) and a high-dose group (tranilast 200mg TID) in this trial to preliminarily evaluate the feasibility of applying tranilast in the clinical treatment of BPH, laying the foundation for new treatment methods for BPH in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign prostatic hyperplasia aged 55 to 75 years old;
* The patient's prostate volume is greater than 40mL;
* There is urinary obstruction, with an International Prostate Symptom Score (IPSS) greater than or equal to 8 points, and a maximum urinary flow rate of less than 15ml/s (urinary flow rate is not measured in patients with indwelling catheters).

Exclusion Criteria:

* Urinary disorders caused by neurogenic diseases;
* Acute urinary tract infections have not been effectively controlled;
* There are factors of lower urinary tract obstruction other than BPH, such as urethral stricture;
* History of radiation therapy or surgery in the lower urinary tract or pelvic cavity;
* Have ever suffered from tumor of urinary system, or suspected of suffering from tumor of urinary system (such as bladder cancer cancer, prostate cancer);
* Current or past liver function abnormalities (exceeding the test reference value limit);
* Abnormal renal function (exceeding the test reference value limit);
* Currently taking warfarin;
* Allergic to tranilast or drug preparations;
* Suffering from other major diseases (malignant tumors, autoimmune diseases, angina pectoris, heart failure, severe respiratory and digestive diseases, etc.), and not yet clinically cured;
* Other researchers believe that patients who are not suitable to participate in this trial.

Ages: 55 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prostate volume | The first month and the sixth month
  No minimum and maximum values, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
International prostate symptom score | The first, third and sixth month
  The minimum value is 0, and maximum values 35. Higher scores mean a worse outcome.
Quality of life score | The first, third and sixth month
  The minimum value is 0, and maximum values 6. Higher scores mean a worse outcome.
International Index of Erectile Function | The first, third and sixth month
  The minimum value is 0, and maximum values 25. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai General Hospital, Shanghai, Outside U.S./Canada
  - Shanghai General Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR